CLINICAL TRIAL: NCT05943379
Title: An Open-label, Single Arm, Single Center Phase 2 Study of RC48-ADC (IV) in Combination With Gemcitabine(Intravesical) in High Risk NMIBC Subjects (BCG Naïve or BCG Unresponsive) That Expresses HER2 (IHC 1+ and Greater)
Brief Title: RC48-ADC in Combination With Gemcitabine in High Risk NMIBC Subjects
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C028
Record Dates: First submitted 2023-03-13; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-05

CONDITIONS: NMIBC
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cohort 1 (Experimental): BCG Naïve
  Interventions: Drug: RC48-ADC in Combination with gemcitabine
- cohort 2 (Experimental): BCG Unresponsive
  Interventions: Drug: RC48-ADC in Combination with gemcitabine

INTERVENTIONS:
Drug: RC48-ADC in Combination with gemcitabine — RC48-ADC IV (intravenous) 2.0mg/kg IV, Q2W, 8W; Q4W, 40W Gemcitabine Intravesical 1000mg induction QW,8W; maintenance Q4W,40W

SUMMARY:
In this study, participants with high risk non-muscle-invasive bladder cancer (NMIBC) who are BCG Naïve or BCG Unresponsive and are considered ineligible for or have refused to undergo radical cystectomy, will receive RC48-ADC in combination with gemcitabine.

DETAILED DESCRIPTION:
The study will be comprised of 2 cohorts. The cohort 1 is BCG Naïve and cohor 2 is BCG Unresponsive.

All participants will receive RC48-ADC(IV) in combination with gemcitabine(intravesical). Treatment on the study will occur during the induction and maintenance phases, and participants will enter a follow-up period after completion of the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent to participate in the study and sign an informed consent form.

2. Male or female, age ≥ 18 years. 3. Disease satisfies.

* Diagnosis in accordance with the Chinese Guidelines for the Treatment of Bladder Cancer (2022) high-risk non-muscle invasive bladder cancer (NMIBC) and meeting any of the following ± carcinoma in situ (CIS): 1. stage T1 tumor of any grade; 2. high-grade tumor; 3. multiple and/or recurrent tumors, with recurrent tumors excluding low-grade solitary tumors.
* Histopathological satisfaction of uroepithelial carcinoma predominant by histopathology, confirming the absence of muscular infiltration.
* Completion of TURBT and resection of all visible lesions within 3 weeks prior to study dosing.
* Clinical staging (cTa/T1±CIS, N0, M0) and absence of distant metastases as assessed by imaging (which needs to include at least CTU) within 3 months prior to enrollment.

  4. 4. Prior BCG treatment.
  1. Cohort 1 is high-risk NMIBC patients who have not received prior BCG therapy: high-risk NMIBC patients who have not received prior BCG therapy due to subjective and objective conditions, including one of the following 1. patient refusal to receive BCG therapy; 2. presence of contraindications to BCG therapy; 3. BCG inaccessibility.
  2. Cohort 2 was high-risk NMIBC patients with BCG non-response, and BCG non-response met any of the following: 1. presence of persistent/recurrent high-risk NMIBC within 12 months (±1 month) of completing adequate BCG therapy; 2. high-grade T1 disease at first assessment after induction phase BCG therapy. Note: Adequate BCG therapy is defined as at least 5 BCG bladder instillations completed within 2 months and at least 2 BCG bladder instillations completed in any 6 consecutive weeks over the next 10 months, i.e., at least "5+2" BCG bladder instillations completed over an approximately 12-month period.

  5. Subjects who have been assessed by a urologist to be unsuitable for radical bladder cancer surgery or who have refused radical bladder cancer surgery.

  6. Subjects whose tumor tissue obtained by TURBT within 3 weeks meets 1+, 2+ or 3+ HER2 expression by immunohistochemistry (IHC) at the study center.

  7. ECOG physical status score of 0-2. 8. Adequate cardiac, bone marrow, liver, and renal function, which should meet the following criteria within 7 days prior to study dosing (normal values are based on the clinical trial center).
* Left ventricular ejection fraction ≥ 50%.
* Hemoglobin ≥ 9 g/dL.
* Absolute neutrophil count (ANC) ≥ 1.5×109/L.
* Platelets ≥ 100×109/L.
* Serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN).
* ALT and AST ≤ 2.5×ULN.
* blood creatinine ≤ 1.5 × ULN or creatinine clearance (CrCl) ≥ 50 mL/min calculated according to the Cockcroft-Gault formula method.

  9. Female subjects should be surgically sterilized, post-menopausal, or agree to use at least one medically approved contraceptive (e.g., IUD, pill, or condom) during study treatment and for 6 months after the end of the study treatment period, and must have a negative blood pregnancy test within 7 days prior to study enrollment; false-positive results may be excluded by the investigator after enrollment. Male subjects should agree to use at least one medically approved contraceptive during the study treatment period and for 6 months after the end of the study treatment period.

  10. be willing and able to comply with the trial and follow-up procedural arrangements.

Exclusion Criteria:

1. muscle-invasive bladder cancer (T2 and above) and/or with regional lymph nodes and distant metastases
2. Combined extra-vesical (i.e. urethral, ureteral or renal pelvis) uroepithelial carcinoma.
3. Received any other antitumor therapy, such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc., within 4 weeks prior to study dosing, excluding 1 dose of infusion chemotherapy completed immediately after TURBT.
4. Have not recovered from an adverse event caused by a previously applied antineoplastic agent to CECAT 5.0 grade 0-1 within 2 weeks prior to the start of study dosing.
5. Those who have undergone major surgery within 4 weeks prior to the start of study dosing or who are scheduled to undergo major surgery during the trial.
6. Serum virological tests (based on the normal values of the study center).

   * Positive HBsAg or HBcAb test result with a positive HBVDNA copy number.
   * Positive HCVAb test result together with a positive HCVRNA test result.
   * Positive HIVAb test result.
7. live vaccine received within 4 weeks prior to the start of study dosing or scheduled to receive any vaccine (except novel coronavirus vaccine) during the study period.
8. heart failure classified as grade 3 or higher by the New York Heart Association (NYHA) of America.
9. the presence of a serious arterial/venous thrombotic event or cardiovascular accident such as deep vein thrombosis, pulmonary embolism, cerebral infarction, cerebral hemorrhage, or myocardial infarction within 6 months prior to study dosing, except for lacunar cerebral infarction that is asymptomatic and does not require clinical intervention
10. the presence of an active infection requiring systemic treatment, such as active tuberculosis
11. the presence of active, unstably controlled systemic disease or serious comorbidity as judged by the investigator, including diabetes mellitus, hypertension, cirrhosis, interstitial pneumonia, obstructive pulmonary disease, complications that could cause the subject to undergo intravesical therapy and/or general anesthesia
12. having any other disease, metabolic abnormality, physical examination abnormality or laboratory test abnormality that, in the judgment of the investigator, gives reason to suspect that the patient has a disease or condition that is inappropriate for the use of the study drug or that will affect the interpretation of the study results, or that places the patient at high risk
13. the presence of an active autoimmune disease requiring systemic therapy (e.g., use of immunomodulatory drugs, corticosteroids, or immunosuppressants) prior to the start of study dosing, allowing for associated replacement therapy (e.g., thyroxine for adrenal or pituitary insufficiency, or replacement therapy with physiologic corticosteroids)
14. other malignancies within 5 years prior to the start of study dosing, with the following exceptions.

    * Malignancies that can be expected to resolve with treatment (including, but not limited to, adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or radical surgically treated ductal carcinoma in situ of the breast).
    * Patients with prostate cancer with prior specific treatment (surgery or radiation therapy).

      1. T2N0M0 or earlier stage.
      2. Gleason score ≤ 7 and prostate-specific antigen (PSA) undetectable for at least 1 year after anti-androgen therapy.
      3. Patients with viable specific therapy or on active surveillance without specific therapy, with stable disease 1 year prior to study entry.
15. previous history of allogeneic HSCT or organ transplantation
16. known hypersensitivity to recombinant humanized anti-HER2 monoclonal antibody-MMAE coupling agent drug and its components or hypersensitivity to gemcitabine and any excipients
17. women who are pregnant or breastfeeding.
18. estimated insufficient patient compliance to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
12-month Disease Free Survival Rate | 12 month

SECONDARY OUTCOMES:
Complete Response Rate | 3 month
6-month Disease Free Survival Rate | 6 month
18-month Disease Free Survival Rate | 18 month
24-month Disease Free Survival Rate | 24 month
Recurrence-free survival | up to 24 months
Progression-Free Survival | up to 24 months
Overall Survival | up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hosptital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No